CLINICAL TRIAL: NCT00334360
Title: Do Dexmedetomidine and Buspirone Synergistically Reduce the Threshold, Gain, and Maximum Intensity of Shivering?
Brief Title: Dexmed/Buspirone Synergism on Shivering
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Dexmed/Buspirone
Record Dates: First submitted 2006-06-06; First posted 2006-06-07 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia | interventions — Dexmedetomidine; Buspirone; Busulfan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): dexmedetomidine
  Interventions: Drug: dexmedetomidine
- 2 (Experimental): Buspirone
  Interventions: Drug: buspirone
- 3 (Experimental): Buspirone and dexmedetomidine
  Interventions: Drug: Bus and Dex
- Control (Placebo Comparator): No drug
  Interventions: Drug: Control

INTERVENTIONS:
Drug: dexmedetomidine — Dexmedetomidine (delivered by a computer-controlled IV infusion to target a plasma concentration of 0.6 ng/mL) will be given during controlled hypothermia
  Arms: 1
Drug: buspirone — Buspirone, 60 mg orally, will be given during controlled hypothermia.
  Arms: 2
Drug: Bus and Dex — the combination of 60 mg buspirone and dexmedetomidine (target plasma concentration of 0.6 ng/mL) will be given during controlled hypothermia
  Arms: 3
Drug: Control — No drugs given during controlled hypothermia
  Arms: Control

SUMMARY:
The purpose of this research is to determine if the combination of buspirone and dexmedetomidine are effective as a treatment to induce therapeutic hypothermia.

The design of the study includes four study days done in random order. The days are as follows: 1) Control (no drug); 2) Buspirone 60 mg orally; 3) Dexmedetomidine (delivered by a computer-controlled IV infusion to a target plasma concentration of 0.6 ng/ml); and, 3) the combination of buspirone 60 mg and dexmedetomidine (target plasma concentration of 0.6 ng/ml). a 20 cm-long catheter will be inserted into a cubital vein using standard aseptic technique In addition to the PIC line catheter, a simple peripheral catheter will be inserted into the other arm for drug administration.

Throughout the study period, mean-skin temperature will be maintained at 31°C by adjusting the temperature of circulating water (Cincinnati Sub-Zero, Cincinnati, OH) and forced-air warmers (Augustine Medical, Inc., Eden Prairie, MN). Furthermore, the back, upper-body, and lower-body will individually be maintained at the designated skin temperature. Lactated Ringer's solution cooled to ≈3°C will be infused via the PIC-line at rates sufficient to decrease tympanic membrane temperature ≈1.5°C/h. Fluid will be administered as long as oxygen consumption or electromyographic intensity (see below) continues to increase or a total of 5 liters of fluid is given. Heart rate will be measured continuously using an electrocardiogram; blood pressure will be determined oscillometrically at 5 min intervals at the ankle. In case heart rate and/or blood pressure changes unexpectedly (by more than 30% of the baseline), the study will stop and the volunteer will be re-warmed immediately.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* normal weight (BMI <35)
* healthy

Exclusion Criteria:

* obese (BMI >35)
* taking any drugs
* thyroid disease, dysautonomia, or Raynaud's syndrome
* severe claustrophobia

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2004-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Shivering threshold | 3 hours
maximum intensity of shivering | 3 hours
gain of shivering | 3 hours

SECONDARY OUTCOMES:
hemodynamic responses | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Lenhardt, MD, PhD, Principal Investigator — University of Louisville School of Medicine
Locations (1):
- Outcomes Research Institute, University of Louisville, Louisville, Kentucky, United States